CLINICAL TRIAL: NCT06413511
Title: A Phase 1b, Dose Escalation, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacological Effect of a Single Intravenous Infusion of Belantamab in Participants With Autoimmune Disease
Brief Title: A Study to Investigate the Safety and Pharmacological Effect of a Single Intravenous Infusion of Belantamab in Male and Female Participants Aged 18 to 75 With Autoimmune Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 221615; 2023-510340-20-00 (Other: EU CT Number)
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Diseases
Keywords: Systemic Lupus Erythematosus; Belantamab (GSK2857914); Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases; Lupus Erythematosus, Systemic | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab (Experimental)
  Interventions: Biological: Belantamab

INTERVENTIONS:
Biological: Belantamab — Belantamab will be administered
  Other Names: GSK2857914

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability profile of belantamab. The study will also assess how the levels of belantamab change over time and body's reaction to it in participants with stable but active autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) from 18 to 40 kilograms per square meter (kg/m^2) (BMI = weight/height^2), inclusive, and body weight of >=40 kilogram (kg)
* IgM >= lower limit of normal (LLN) (40 milligram per deciliter [mg/dL]) at initial screening visit (ISV)

Participants with systemic lupus erythematosus (SLE) must also meet the following inclusion criteria:

* Documented clinical diagnosis of SLE according to the European League Against Rheumatism (EULAR) or American College of Rheumatology (ACR) Classification Criteria
* Positive anti-double stranded deoxyribonucleic acid (anti-dsDNA) autoantibody and/or positive antinuclear antibody (ANA) test results, using central lab test, at ISV.
* SLE Disease Activity Index 2000 (SLEDAI-2K) total score of >=6 at ISV.
* Failure to adequately respond to at least two immunosuppressive therapies.

Participants with Rheumatoid Arthritis (RA) must also meet the following inclusion Criteria:

* Meets ACR/EULAR 2010 RA Classification Criteria with a duration of RA disease of >=6 months at time of ISV
* Positive rheumatoid factor (RF) and/or anti-cyclic citrullinated peptide (anti-CCP) test results, using central lab test, at ISV.
* Have moderate to severe active disease as defined by >=3/68 Tender and >=3/66 Swollen joint count at ISV and Baseline.
* Failure to adequately respond to at least two immunosuppressive therapies.

Participants with antiphospholipid syndrome (APS) must also meet the following inclusion criteria:

* Documented diagnosis of APS meeting the 2023 ACR/EULAR APS classification criteria
* Positive lupus anticoagulant test or moderate to high titers of positive IgG/IgM anticardiolipin (aCL) or moderate to high titers of IgG/IgM anti-beta2-glycoprotein I antibody using central lab test, at ISV
* Clinical features attributable to antiphospholipid antibodies that are resistant to warfarin and/or heparin:

  * Thrombotic event within last 18 months despite adequate anti-coagulation therapy and/or
  * Persistent thrombocytopenia and/or
  * Persistent autoimmune hemolytic anemia
* Sex and Contraceptive /Barrier requirements for females.

Exclusion criteria:

SLE specific exclusion:

* Any acute, severe lupus related flare during the Screening Period that needs immediate treatment
* Has any unstable or progressive manifestation of SLE
* Significant, likely irreversible organ damage related to SLE

RA specific exclusions:

* RA functional status class IV according to the ACR 1991 revised criteria
* Adult Juvenile RA

APS specific exclusions:

* Acute thrombosis (arterial or venous acute thrombosis diagnosis) less than 30 days before study ISV
* Catastrophic APS classification within the prior 90 days of ISV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Up to Week 12
Number of participants with clinically important findings in vital signs | Up to Week 12
Number of participants with clinically important findings in electrocardiogram | Up to Week 12
Number of participants with clinically important findings in echocardiogram | Up to Week 12
Number of participants with clinically important findings in hematology | Up to Week 12
Number of participants with clinically important findings in clinical chemistry | Up to Week 12
Number of participants with clinically important findings in urinalysis parameters | Up to Week 12
Number of participants with clinically important finding in corneal toxicity | Up to Week 12

SECONDARY OUTCOMES:
Change from Baseline in Immunoglobulin (Ig) M (IgM) | Baseline (Day 1) and up to Week 12
Area under the concentration-time curve from time 0 to the last quantifiable concentration [AUC(0-t)] of belantamab | Up to 12 weeks
Area under the concentration-time curve from time 0 to infinity [AUC(0-inf)] of belantamab | Up to 12 weeks
Maximum observed plasma drug concentration [Cmax] of belantamab | Up to 12 weeks
Number of participants with Anti-Drug Antibodies (ADAs) against belantamab | Up to 12 weeks
Titers of ADAs against belantamab | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/